CLINICAL TRIAL: NCT05249179
Title: Comparison of the Effects of Oral Stimulation and Non-nutritive Sucking Practices on the Transition to Full Oral Feeding in Infants With a Gestational Age of 26-32 Weeks
Brief Title: Comparison of the Effects of Oral Stimulation and Non-nutritive Sucking Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E2-21-883
Record Dates: First submitted 2021-12-11; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Premature; Nutrition Disorders; Sucking Behavior
Keywords: Sucking; Oral stimulation; Premature baby
MeSH Terms: conditions — Premature Birth; Nutrition Disorders; Sucking Behavior | interventions — Pacifiers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Oral stimulation) (Experimental): The group that will receive oral stimulation with the Backman method once a day from the 29th week
  Interventions: Other: Oral stimulation
- Group 2 (Pacifier) (Experimental): The group that will be given a pacifier three times a day from the 29th week
  Interventions: Other: Pacifier
- Group 3 (oral stimulation + pacifier) (Experimental): Starting from the 29th week, the group will be given a pacifier three times a day and a Backman oral stimulation will be applied once a day.
  Interventions: Other: Pacifier; Other: Oral stimulation
- Group 4 (Enteral feeding by tube) (No Intervention): The group fed enterally by tube in routine practice, in which no intervention will be made.

INTERVENTIONS:
Other: Pacifier — Preterm infants in Groups 2 and 3 will suck a pacifier 3 times a day (09:00, 12:00, 15:00) for 3 minutes before feeding and then they will be fed with the O/G feeding tube.
  Arms: Group 2 (Pacifier); Group 3 (oral stimulation + pacifier)
Other: Oral stimulation — Infants in groups 1 and 3 will receive a prefeeding oral stimulation program once a day, 15 to 30 minutes before a tube feeding. Oral stimulation programs will be delivered by trained nurses or pediatric physical therapies. Nurses will be trained to deliver the stimulation program to the infants, by a member from the pediatric physical therapies medical staff, before the beginning of the study. Based on Backman's principles, the pre-feeding oral stimulation program consisted of a 12-minute stimulation program that included stroking the cheeks, lips, gums, and tongue.
  Arms: Group 1 (Oral stimulation); Group 3 (oral stimulation + pacifier)

SUMMARY:
This study, it was aimed to compare the effects of oral stimulation and non-nutritive sucking practices on the transition to full oral feeding in babies with a gestational age of 26-32 weeks. Non-oral feeding methods are frequently used in babies born prematurely since sucking and sucking-swallowing coordination have not yet developed. While some premature babies gain the sucking and swallowing reflexes faster, some of them cannot develop this reflex for a long time, so the length of hospital stay is prolonged. All infants who can be fed completely enterally (PMA >29 weeks) will be randomized into 4 groups as oral stimulation (group 1), pacifier (group 2), oral stimulation + pacifier (group 3), and control group by using a stratified blocked randomization method with a block size of 4. Stratification on GA (26-27, 28-29, 30-32 weeks GA) was used to ensure that the groups had similar gestational age distribution. The time of the patients to start breastfeeding and the length of hospital stay (days) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies born between 26-32 weeks (including 26 and 32 weeks)

Exclusion Criteria:

* Babies with congenital anomalies
* Babies born with asphyxia
* Babies with major GIS anomalies
* Babies who have undergone major GIS surgery

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Full oral feeding time (postmenstruel week) | 2 years
  The effect of oral stimulation and/or pacifier use on full oral feeding time in premature infants.
Hospital stay (days) | 2 years
  The effect of oral stimulation and/or pacifier use on hospital stay in premature infants

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Altuntas, Proff, Study Director — Ankara Bilkent Central Hospital, Neonatal Unit; Suna S Oguz, Proff, Study Director — Ankara Bilkent Central Hospital, Neonatal Unit; Mustafa S Akin, Specialist, Study Director — Ankara Bilkent Central Hospital, Neonatal Unit

IPD SHARING:
Plan to Share IPD: Undecided
No agreement yet to share with other researchers